CLINICAL TRIAL: NCT06737640
Title: Evaluation of Biochimical, Bioumoral and Molecular Features as Predicitive Factors of Response or Toxicities During Immunotherapy Treatment of Uterine Cancer Patients
Brief Title: Evaluation of Clinical and Molecular Biomarkers in Immunotherapy Treatment in Gynecologic Cancer
Acronym: Immuno-Gyn
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6881
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Cervical Cancer; Endometrial Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Immunotherapy has changed the therapeutic approach for gynecologic gynecological malignancies such us endometrial and cervical cancer. Despite literature data support the strong effect of immunotherapy in these cancers, a share of patients do not respond to immunotherapy. Furthermore the extremely variable immune-related spectrum of toxicity in terms of events and timing makes it necessary to identify predictive factors for the development of these side effects.

Hyphotesis: To evaluate the presence of biochemical, bioumoral and or molecular predictive factors in patients affected by endometrial and cervical cancer treated with immunotherapy plus chemotherapy, immunotherapy plus tyrosine kinase inhibitors (TKI) or immunotherapy alone.

Methodology: We will retrospectively collect data about patients affected by advanced, recurrent or metastatic endometrial cancer (EC) and recurrent cervical cancer (CC) treated with immunotherapy.

We will investigate whether there is a statistically significant difference in the efficacy of immunotherapy according to biochemical, biohumoral and or molecular factors and survival outcomes. Moreover, we will evaluate whether there is a correlation between biochemical, biohumoral and or molecular factors and immune-related adverse events (irAE).

ELIGIBILITY:
Inclusion Criteria:

* Females aged ≥ 18 years at the time of inclusion in the study.
* Patients diagnosed with advanced, metastatic or recurrent endometrial and cervical cancer treated at the Fondazione Policlinico Universitario Agostino Gemelli IRCCS.
* Patients with histological confirmation of endometrial and cervical cancer, according to the histotypes suitable for immunotherapy.
* Patients previously treated under Nominal Use and/or Expanded Access Program (EAP) programs can be enrolled in the study.
* Patients who have received at least 1 dose of immunotherapy after starting treatment.
* Signature of the informed consent or declaration in lieu of the consent form where applicable

Exclusion Criteria:

* Use of immunotherapy within an experimental protocol.
* Patients who continued therapy at another center.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced, metastatic or recurrent endometrial cancer and advanced, metastatic or recurrent cervical cancer undergoing treatment with immunotherapy in combination with chemotherapy or tyrosine kinase inhibitors or with immunotherapy as monotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-12-16 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of biomarkers in immunotherapy in endometrial cancer. | 12 months
  Evaluate the association between biochemical, biohumoral and molecular factors and survival outcome in patients with advanced, metastatic or recurrent endometrial cancer treated with immunotherapy and chemotherapy, immunotherapy and tyrosine kinase inhibitors or immunotherapy in monotherapy.
Evaluation of biomarkers in immunotherapy in cervical cancer. | 12 months
  Evaluate the association between biochemical, biohumoral and molecular factors and survival outcome in patients with advanced, metastatic or recurrent cervical cancer treated with immunotherapy and chemotherapy, immunotherapy and tyrosine kinase inhibitors or immunotherapy in monotherapy.

SECONDARY OUTCOMES:
Evaluation of immuno-related adverse events (irAEs) in gynecologic cancer. | 12 months
  Evaluate the association between biochemical, biohumoral and possibly molecular factors and the onset of immune-related adverse events during and after the end of immunotherapy treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Eleonora Palluzzi, MD, Principal Investigator — Fondazione Policlinico Agostino Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli, IRCCS, UOC Ginecologia Oncologica, Rome, Lazio, Italy